CLINICAL TRIAL: NCT04170426
Title: Phase 1/2a Clinical Study for Subjects With Rheumatoid Arthritis (RA) Using Multiple Dose Intravenous Infusions of Autologous Adipose Tissue-Derived Mesenchymal Stem Cells (AdMSCs)
Brief Title: Autologous Adipose-derived Stem Cells (AdMSCs) for Rheumatoid Arthritis
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celltex Therapeutics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTX0019-001
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Combined Phase 1 dose escalation study and Phase 2a randomized, placebo controlled and double blinded study using autologous adipose stem cells (Celltex AdMSCs) for rheumatoid arthritis patients who failed disease-modifying antirheumatic drug (DMARDs).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1 ARM 0 (Experimental): 9 subjects receive dose escalation of autologous AdMSCs via Intravenous infusion in Phase 1
  Interventions: Biological: autologous adipose derived stem cells
- Phase 2 ARM 1 (Active Comparator): 30 subjects receive three doses of 2.0-2.86×10^6 cells/kg on day 1, 4 and 7 via Intravenous infusion in Phase 2a
  Interventions: Biological: autologous adipose derived stem cells
- Phase 2 ARM 2 (Placebo Comparator): 15 subjects receive three doses of placebo on day 1, 4 and 7 via Intravenous infusion in Phase 2a
  Interventions: Biological: autologous adipose derived stem cells

INTERVENTIONS:
Biological: autologous adipose derived stem cells — Culture expanded mesenchymal stem cells isolated from patient's own abdominal fat tissue
  Other Names: Celltex-AdMSCs

SUMMARY:
This is an investigational new drug clinical trial for combined Phase 1 dose escalation study and Phase 2a randomized, placebo controlled and double blinded study using intravenous injection of autologous adipose stem cells (Celltex AdMSCs) for rheumatoid arthritis patients. All subjects are monitored for safety (adverse events/severe adverse events) and evaluated for RAPID3, DAS28 and ACR20 regarding AdMSCs up to 52 weeks study duration.

ELIGIBILITY:
Inclusion Criteria:

* Must pass communicable disease screen tests for HIV, syphilis, Hepatitis B and C Consistent with American Rheumatism Association-European League Against Rheumatism (ACR/EULAR) 2010 rheumatoid arthritis classification criteria
* Active Rheumatoid Arthritis, see RA functional status of class I-IV
* Patients must meet at least one of the following: > 6 swollen joints and ≥ 6 involved joints (tenderness, swelling, deformity, pain on motion, or decreased motion) and morning stiffness ≥ 45 minutes based on 68 joint count.
* Patients must also meet at least one of the following: rheumatoid factor (RF) > 15 IU/mL or > 1:16, C-reactive protein (CRP) > 2.0 mg/dL, Erythrocyte Sedimentation Rate (ESR) > 30 mm/hour, and anti-cyclic citrullinated protein (Anti-CCP) > 20 U/mL, TNFα > 2.8 pg/mL.
* Patients must have failed anti-rheumatoid drug due to adverse event or inefficacy for at least 12 week and at least 4 weeks on stable dose of methotrexate ≤ 25 mg/week, or leflunomide ≤ 20 mg/day, or sulfasalazine ≤ 3 g/day, or steroids (Prednisone <10 mg/day).
* For other medications, patients must be on the stable dose for at least 4 weeks prior to study entry in order to preclude changes to patient medication while participating on the study to ensure that a medication change could become a confounding factor in data interpretation.
* All patients must be clinically stable with no significant changes in health status a minimum of at least 4 weeks prior to randomization and confirming patient eligibility

Exclusion Criteria:

1. Current or prior to treatment

   * Participation in another clinical study (with use of another Investigational Medical Product) within 3 months prior to study treatment start
   * Evidence of immune suppression related to prior/current therapy
   * > 10% change in delivered monthly dose of anti-rheumatoid medications within 4 weeks prior to this stem cell infusion
   * Use of a new or additional anti-rheumatoid medication within 6 weeks prior to this stem cell infusion
   * Use of other stem cell therapy within 12 weeks prior to this stem cell therapy
   * Unwillingness or inability to comply with study procedures
2. Concurrent Conditions

   * Clinically active malignant disease
   * Severe bladder or thrombotic disorder
   * History of known pulmonary embolism or known secondary anti-phospholipid syndrome
   * Known or suspected hypersensitivity to any components used to culture or store the AdMSCs, e.g. sulfur or sulfonamide
   * Known or suspected antibodies to any components used to culture the AdMSCs, e.g. BSA and sulfur containing products (e.g., DMSO)
   * Active infection at time of planned study treatment start
   * Age related pathology likely to inhibit study participation or completion
   * Major trauma or surgery within 14 days of study treatment start
   * Mental condition rendering the subject (or the subject's legally acceptable representative[s]) unable to understand the nature, scope and possible consequences of the study
   * Alcohol, drug, or medication abuse within one year before study treatment start
   * Any condition that, in the Investigator's opinion, is likely to interfere with evaluation of the AdMSC therapy or satisfactory conduct of the study
   * Irreversible severe end organ failure, such as heart failure/attack, stroke, liver and renal failure
   * Heavy smokers, bed-bound patients, patients or family history with hypercoagulable status, such as protein C/protein S deficiency, factor V Leiden, prothrombin gene mutation, dysfibrinogenemia, etc.
3. Laboratory Parameters

   * Hepatic impairment, defined as any of ALT, AST, LDH or bilirubin > 2 x the upper limit of normal (ULN) range according to local laboratory standards
   * Renal impairment, defined as serum creatinine > 133 mmol/L (1.5 mg/dL)
   * Positive virology/serology for human immunodeficiency virus (HIV), hepatitis B (HBsAg positive), hepatitis C and/or syphilis
4. Pregnancy / contraception

   * Pregnant, breastfeeding, or desire to become pregnant or unwilling to practice birth control during participation in the study duration, unless surgically sterilized or postmenopausal during the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Events and Sever Adverse Events | 52 weeks
  The total number of adverse events and severe adverse events related and non-related with AdMSCs will be recorded to indicate the safety and tolerability.

SECONDARY OUTCOMES:
Efficacy of Celltex AdMSCs | 52 weeks
  Proportion of ACR 20 patients (swollen joints, tender joints, patient assessment of pain, RAPID3, DAS28-CRP and blood inflammatory panel tests) in comparison between baseline and post-treatment follow-up data.

CONTACTS AND LOCATIONS:
Overall Officials: Derek W Guillory, MD, Principal Investigator — Root Causes Medicine

IPD SHARING:
Plan to Share IPD: No